CLINICAL TRIAL: NCT00164684
Title: Men of Color Fatherhood Education and Violence Prevention Project
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joanne Klevens (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Joanne Klevens, epidemiologist, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCIPC-US4CCU119008051; US4/CCU119008-05-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Spouse Abuse
Keywords: batterers; prevention; African American; Latino

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Father Friendly Initiative

SUMMARY:
A 16 session curriculum, developed for noncustodial African American and Latino fathers to improve knowledge, attitudes and skills and enable participants to remain non-violent towards their partners will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Noncustodial fathers
* African American or Latino
* At high risk for violence (prior perpetration, un/underemployment)

Exclusion Criteria:

* Substance abusers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rich, MD, Principal Investigator — Boston Public Health Commission
Locations (1):
- Boston Public Health Commission, Boston, Massachusetts, United States